CLINICAL TRIAL: NCT03197285
Title: Effectiveness of an Eye-Cervical Re-education Program (ECRP) to Decrease Pain and Increase Mobility in the Cervical Area Compared to a Combined Physiotherapy Protocol (CPP) in Patients With Chronic Neck Pain Symptoms.
Brief Title: Effectiveness of an Eye-Cervical Re-education Program in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Veronica Perez Cabezas, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U-Cadiz-V Perez-Cabezas
Record Dates: First submitted 2017-06-12; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Neck Pain; Eye Strain
Keywords: neck pain; eye; propioception; range of motion; pain
MeSH Terms: conditions — Neck Pain; Asthenopia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): All patients are given a Combined Physiotherapy Protocol (CPP) consisting of: Thermotherapy (70 w continuous microwave for 10 minutes), therapeutic massage (surface rubbing for 5 minutes, 10 minutes of compression and kneading massage and 2 minutes of final surface friction), application of analgesic currents (TENS, by self-adhesive silicone electrodes 4x4 cm, symmetrical biphasic rectangular current, 200 µs width pulse, a frequency of 1 Hz for 10 minutes. The patient should notice a slight vibration, without it being painful).
  Interventions: Other: Combined Physiotherapy Protocol
- Experimental Group (Experimental): All patients are given a Combined Physiotherapy Protocol (CPP) consisting of: Thermotherapy (70 w continuous microwave for 10 minutes), therapeutic massage (surface rubbing for 5 minutes, 10 minutes of compression and kneading massage and 2 minutes of final surface friction), application of analgesic currents (TENS, by self-adhesive silicone electrodes 4x4 cm, symmetrical biphasic rectangular current, 200 µs width pulse, a frequency of 1 Hz for 10 minutes. The patient should notice a slight vibration, without it being painful). The ECRP developed by Revel et al.(Revel et al., 1994) was also applied to patients in the experimental group.
  EYE-CERVICAL RE-EDUCATION PROGRAM (ECRP) This includes a total of 10 exercises that has proprioceptive reprogramming in the cervical area
  Interventions: Other: EYE-CERVICAL RE-EDUCATION PROGRAM

INTERVENTIONS:
Other: EYE-CERVICAL RE-EDUCATION PROGRAM — Subjects received a total of ten sessions on alternate days.
  This includes a total of 10 exercises that has proprioceptive reprogramming in the cervical area with the following phases:
  1. To stimulate ocular mobility without including the cervical movement. The patient was placed in the supine position and the physiotherapist seated, at the height of the head.
  2. To exercise cervical mobility with restricted eye movement. The patient is placed on a rotating stool. The ocular mobility is excluded with opaque glasses that allowed exclusively the foveal vision
  3. Finally we stimulate eye and neck movement coordination. The patient continued to sit on the stool, this time without the glasses.
  Arms: Experimental Group
Other: Combined Physiotherapy Protocol — Thermotherapy (70 w continuous microwave for 10 minutes), therapeutic massage (surface rubbing for 5 minutes, 10 minutes of compression and kneading massage and 2 minutes of final surface friction), application of analgesic currents (TENS, by self-adhesive silicone electrodes 4x4 cm, symmetrical biphasic rectangular current, 200 µs width pulse, a frequency of 1 Hz for 10 minutes. The patient should notice a slight vibration, without it being painful).
  Arms: Control Group

SUMMARY:
The aim of the present study is to value the effectiveness of an Eye-Cervical Re-education Program (ECRP) to decrease pain and increase mobility in the cervical area compared to a Combined Physiotherapy Protocol (CPP) in patients with chronic neck pain symptoms.

DETAILED DESCRIPTION:
Background:

In Physiotherapy there is a growing interest of authors to clarify the relationship between the visual system and the neck. Aspects such as deficiencies in eye movement during cervical rotation are common disorders in patients who have suffered whiplash trauma or have dizzy syndromes. On the other hand, deep muscle disorders of the neck are related to the decrease in cervical-ocular reflex. Furthermore, some disorders in eye movements in patients with idiopathic neck pain have been identified.

Consequently, a pragmatic approach to multimodal intervention has been recommended to address changes in sensorimotor control at the cervical level. For this purpose, head-neck sensitization exercises (joint position sense training with head relocation), oculo-motor exercises (ie, eye stability, eye-neck coordination) or balance training have been proposed. These programs lead to a sensorimotor control, reducing pain and disability in the neck. However, it is not known if this approach to treatment is a significant improvement when compared to the implementation of other physiotherapy procedures, so it is unknown if the application of training oculocervical proprioception is more advisable than other modalities of physiotherapy treatment for the improvement of CNP symptoms.

Material and method:

This research is an analytical, longitudinal, prospective, experimental, evaluator blinded study. It is controlled with two parallel groups, randomized clinical trial.

The sample consisted of patients recruited in a Physiotherapy consultation in Cadiz (Spain). These assessments were made before and after the start of program and to the end of intervention (8 months).

Patients were randomized to control or experimental group. All patients are given a Combined Physiotherapy Protocol, no apply an Eye-Cervical Re-education Program in subjects in the first group and performing an Eye-Cervical Re-education Program in the second. This program was carried out by the physiotherapist. Subjects received a total of ten sessions on alternate days.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: to show symptoms and clinical signs of neck pain, have a medical diagnosis, meet the following lines according to the classification proposed by the Working Group "Bone and Joint Decade 2000-2010" (Axis 1:Health problem receiving health care, Axis II: tertiary care; healthcare in a private Physiotherapy center, Axis III: Grades I and II, Axis IV: Long term, more than three months, Line V: isolated, periodic or permanent Crises) and cervical pain of a mechanical origin, due to repetitive motion or maintenance of positions for long periods.

Exclusion Criteria:

* Dizziness syndrome, microwave contraindications and analgesic currents (therapeutic procedures used), post-traumatic, rheumatologic, neurological, infectious or tumor cervical pain.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change of pain | Baseline and end of treatment(4 weeks)
  Algometer in 6 points (two trapezius, two in angular of the scapula and two sub-occipital)
Change of range of motion | Baseline and end of treatment (4 weeks)
  Measured with inclinometer

SECONDARY OUTCOMES:
Pain Rating Index | Baseline and end of treatment(4 weeks)
  McGill questionnaire in Spanish version
Numerical rating scale for pain | Baseline and end of treatment(4 weeks)
  VAS visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing and Physiotherapy. University of Cadiz, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen LL, Hansen K, Mortensen OS, Zebis MK. Prevalence and anatomical location of muscle tenderness in adults with nonspecific neck/shoulder pain. BMC Musculoskelet Disord. 2011 Jul 22;12:169. doi: 10.1186/1471-2474-12-169. PMID 21777478
- [Background] Treleaven J, Jull G, LowChoy N. Smooth pursuit neck torsion test in whiplash-associated disorders: relationship to self-reports of neck pain and disability, dizziness and anxiety. J Rehabil Med. 2005 Jul;37(4):219-23. doi: 10.1080/16501970410024299. PMID 16024477
- [Background] Revel M, Minguet M, Gregoy P, Vaillant J, Manuel JL. Changes in cervicocephalic kinesthesia after a proprioceptive rehabilitation program in patients with neck pain: a randomized controlled study. Arch Phys Med Rehabil. 1994 Aug;75(8):895-9. doi: 10.1016/0003-9993(94)90115-5. PMID 8053797
- [Background] Treleaven J, Takasaki H. Characteristics of visual disturbances reported by subjects with neck pain. Man Ther. 2014 Jun;19(3):203-7. doi: 10.1016/j.math.2014.01.005. Epub 2014 Jan 27. PMID 24521926
- [Derived] Perez-Cabezas V, Ruiz-Molinero C, Jimenez-Rejano JJ, Chamorro-Moriana G, Gonzalez-Medina G, Chillon-Martinez R. Effectiveness of an Eye-Cervical Re-Education Program in Chronic Neck Pain: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2020 Feb 26;2020:2760413. doi: 10.1155/2020/2760413. eCollection 2020. PMID 32184889